CLINICAL TRIAL: NCT06591780
Title: Innovative Multi-Variable Biofeedback for Improving Gait Performance in Individuals With Diabetic Peripheral Neuropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Institute for Human and Machine Cognition (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Nicole Rendos, Research Scientist, Florida Institute for Human and Machine Cognition
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-2025-0002.1; P30DK111024 (NIH)
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Peripheral Neuropathy; Diabetes Mellitus
Keywords: anterior ground reaction force; biofeedback-induced changes in plantar pressure; diabetic peripheral neuropathy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Real-Time Biofeedback Walking Trials (Experimental): Real-time biofeedback of propulsion and plantar pressure to measure the immediate effects of biofeedback on walking function and gait mechanics.
  Permuted block randomization (blocks of 4) will be used to allocate the order of the biofeedback stimulus (plantar pressure-intervention A or propulsion-intervention B).
  Participants will receive both interventions in session 3, but the order will be randomized.
  Interventions: Other: Clinical Evaluation; Other: Plantar Pressure Biofeedback Gait Training; Other: Propulsion Biofeedback Gait Training

INTERVENTIONS:
Other: Clinical Evaluation — A clinical evaluation occurs at the first study session. The clinical evaluation assesses walking function and mobility, lower extremity, sensation, health-related quality of life (HRQoL) and foot function.
  Session 2 will be a dynamometer-based evaluation of passive ankle stiffness and a 3-dimensional gait analysis to evaluate baseline biomechanics. During Session 3, real-time biofeedback conditions will be used to measure the immediate effects on walking function.
Other: Plantar Pressure Biofeedback Gait Training — Participants will complete a 3-dimensional gait evaluation prior to training, after a 6-minute control bout without biofeedback, and following three 6-minute biofeedback training bouts (total 18-minutes). Individualized biofeedback targets will be calculated from each participant's immediate biofeedback session to best minimize plantar pressure whilst maintaining or enhancing propulsion. Audio-visual biofeedback is provided using a screen placed in front of the treadmill and a speaker. For plantar pressure biofeedback, a visual display of a foot with a colored heat map represents the current plantar pressure, in addition to bar graphs representing real-time movement of plantar pressure in specific areas of the foot. A target is provided using the heat map colors of red and target line on the bar graph. Participants are informed that the target is a measurement of the pressure under their foot, and their goal is to decrease pressure to achieve their target
  Other Names: Intervention A
Other: Propulsion Biofeedback Gait Training — Participants will complete a 3-dimensional gait evaluation prior to training, after a 6-minute control bout without biofeedback, and following three 6-minute biofeedback training bouts (total 18-minutes). Individualized biofeedback targets will be calculated from each participant's immediate biofeedback session to best minimize plantar pressure whilst maintaining or enhancing propulsion. Audio-visual biofeedback is provided using a screen placed in front of the treadmill and a speaker. For propulsion biofeedback, a visual display with a marker represents the current propulsion (peak AGRF) and a target provided to modulate propulsion. Participants are informed that the marker is a measurement of how hard they are pushing the ground backward, and their goal is to push-off more to achieve their target.
  Other Names: Intervention B

SUMMARY:
This study aims to collect data to improve gait function in individuals with Diabetic Peripheral Neuropathy (DPN).

The primary goals are to evaluate:

* Biomechanical mechanisms contributing to abnormal plantar pressure and propulsion during gait in individuals with DPN
* Biofeedback-induced changes in plantar pressure, propulsion, and biomechanics during gait in individuals with DPN

The participants will be required to complete

* Questionnaires
* Clinical examination
* 3-Dimensional gait analysis on an instrumented treadmill
* Visual and auditory biofeedback on the participant's propulsion and plantar pressure metrics provided by a projector screen during walking

DETAILED DESCRIPTION:
Over 38 million adults in the United States (~1 in 7) are living with Diabetes Mellitus (DM), of which diabetic peripheral neuropathy (DPN) is the most common complication, affecting more than 50% of individuals with DM. DPN causes both sensory and motor impairments of the foot and ankle, leading to reduced functional mobility and increased ulceration and amputation risk. Propulsion and plantar pressure are two key interrelated gait parameters contributing to walking function and ulceration risk, respectively. Real-time biofeedback is a non-invasive rehabilitation strategy with significant promise for targeting gait impairments by providing the user with quantitative information regarding a targeted performance variable.

In this study, the team will evaluate multi-joint lower extremity biomechanical responses to univariate propulsion and plantar pressure biofeedback. Secondly, the team will use identified biomechanical compensations to propulsion and plantar pressure biofeedback to develop a multi-variable, implicit, individualized visual biofeedback program to improve gait function in individuals with DPN. Insights into the biomechanical mechanisms underlying plantar pressure and propulsion in people with DPN will allow us to design more informed and effective gait rehabilitation interventions aimed at preventing deleterious outcomes such as ulceration and amputation that can be tailored to individual patient characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Able to walk 10-meters independently without an assistive device
* Sufficient cardiovascular and musculoskeletal health to walk on a treadmill for 6 minutes at a self-selected speed
* Diagnosis of diabetes mellitus
* Diagnosis of diabetic peripheral neuropathy by a physician
* Foot examination within the past 6 months documenting ambulatory status
* Physician clearance

Exclusion Criteria:

* History of amputation
* Active ulceration
* Medial column deformity
* Severe cognitive impairment (MoCA < 10)
* Severe visual impairment
* History of Charcot osteoarthropathy
* History of posterior muscle group lengthening
* History of lower extremity joint replacement
* History of lower extremity and/or foot surgery affecting walking mechanics
* Orthopaedic problems of the lower limbs or spine due to other medical conditions (not diabetes or DPN) that limit walking or cause pain during walking
* Improper footwear for walking and community ambulation
* Cardiovascular or medical condition affecting ability to walk safely
* History of unexplained dizziness or fainting in the past 2 months
* Allergy to adhesive tape or rubbing alcohol

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Biomechanical plantar pressure | Study Session 2 (occurs 24 hours up to 2 weeks after Session 2)
  Plantar pressure is calculated in kilopascals (kPa) using a force sensor placed between the participant's foot and insole of their shoe. The peak plantar pressure in regions of interest (forefoot) will be calculated.
Biomechanical Propulsion | Study Session 2 (occurs 24 hours up to 2 weeks after Session 2)
  Propulsion is calculated as the maximum anteriorly directed ground reaction force during the stance phase of gait using the instrumented (force plate) treadmill.

SECONDARY OUTCOMES:
Changes induced by biofeedback in plantar pressure | Study Session 3 (occurs 24 hours up to 2 weeks after Session 3)
  Plantar pressure measurements will be recorded using insoles placed between the surface of the foot and the insole of the participant's shoe. Marker data, GRFs, and plantar pressure data will be synchronized.
Changes induced by biofeedback in propulsion | Study Session 3 (occurs 24 hours up to 2 weeks after Session 3)
  Ground reaction force (GRF) data will be collected independently from each leg using a split-belt treadmill instrumented with two 6-degree of freedom force platforms. The antero-posterior GRFs (AGRF) will be used to compute propulsion.
Changes induced by biofeedback in biomechanics during gait | Study Session 3 (occurs 24 hours up to 2 weeks after Session 3)
  Lower extremity kinetics and kinematics will be measured using a three-dimensional motion analysis system and split-belt instrumented treadmill. Kinetics and kinematics of the ankle, knee, and hip will be analyzed during gait.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole K Rendos, PhD, Principal Investigator — Florida Institute for Human and Machine Cognition
Locations (1):
- Florida Institute for Human and Machine Cognition, Pensacola, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Data on demographics, medical history, clinical evaluation, questionnaires, walking biomechanics, and plantar pressure data will be collected from individuals (N = 25) with diabetic peripheral neuropathy. Subject-level de-identified data will be preserved and shared in raw and pre-processed forms in ".csv" and ".xlsx" format. Biomechanics data will be processed and saved in ".c3d" formatted files as per standard practice in the field of biomechanics.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All data will be deposited 6 months following the completion of the study. At a minimum, the data will be made available for 3 years after the completion of the study.
Access Criteria: Raw and pre-processed data will be archived through the National Institute of Child Health and Human Development (NICHD) Data and Specimen Hub (DASH). Processed biomechanics data will be archived through SimTK. The archived data will be assigned digital object identifiers (DOI). Both NICHD DASH and SimTK are made available through web-accessible repositories at no cost to users.